CLINICAL TRIAL: NCT05467397
Title: Feasibility Study of [11C]Acetate Positron Emission Tomography (PET) as an Indicator of Early Response to Rapamycin in Lymphangioleiomyomatosis (LAM) Patients
Brief Title: Feasibility of [11C]Acetate-PET in LAM and TSC
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Carmen Priolo, M.D., Ph.D., Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019p003557
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Lymphangioleiomyomatosis; Tuberous Sclerosis Complex
MeSH Terms: conditions — Lymphangioleiomyomatosis; Tuberous Sclerosis | interventions — carbon-11 acetate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients will undergo [11C]acetate PET/CT (Experimental): Patients will undergo a single [11c]acetate PET scan OR Patients will undergo an [11c]acetate PET scan, initiate treatment with rapamycin or rapalogs and receive a second [11c]acetate PET scan 3 or 4 months after starting the treatment.
  Interventions: Drug: [11C]acetate

INTERVENTIONS:
Drug: [11C]acetate — Positron Emission Tomography (PET)
  Other Names: diagnostic test

SUMMARY:
This study aims to assess [11C]acetate positron emission tomography (PET)/computed tomography (CT) as a biomarker for renal angiomyolipomas and pulmonary lymphangioleiomyomatosis (LAM) and an early biomarker of response to rapamycin in LAM patients.

[11C]Acetate is a radioactive form of acetate, a nutrient commonly processed in our body's cells to generate fat and energy. Preclinical studies support the hypothesis that TSC tumors enhance lipid synthesis compared to normal tissues, suggesting that quantification of [11C]acetate in these tumors by PET/CT may provide a metabolic biomarker of disease.

Participants in the study will undergo 1 or 2 PET/CT scans over 3 to 6 months at the Massachusetts General Hospital (Boston, MA). [11C]acetate is administered through an intravenous catheter. This small amount of radioactivity is short-lived and eliminated from the body within a few hours.

DETAILED DESCRIPTION:
Lymphangioleiomyomatosis (LAM) is a rare, multisystem disease of women, consisting of a diffuse proliferation of smooth muscle actin-positive cells (LAM cells), which harbor inactivating mutations in either the TSC1 or TSC2 tumor suppressor gene. These inactivating mutations result in constitutive activation of mammalian/mechanistic TOR (target of rapamycin) complex 1 (mTORC1), which integrates growth factor and nutrient signaling to stimulate cell growth and metabolism. Pulmonary LAM is characterized by associated progressive cystic destruction of the lung parenchyma, recurrent pneumothorax, and chylous pleural effusions. Extrapulmonary proliferative lesions of LAM include renal angiomyolipomas and lymphangiomyomas. LAM can occur as a sporadic disorder where LAM cells harbor somatic inactivating mutations of the TSC1 or TSC2 gene, or in women with Tuberous Sclerosis Complex (TSC).

Rapamycin is an FKBP12-dependent allosteric inhibitor of mTORC1 approved by the FDA for the treatment of LAM and TSC-associated renal angiomyolipomas. Clinical trials of TSC and LAM have shown that 12 month-treatment with rapamycin induces response of renal angiomyolipomas and stabilization of pulmonary function. However, lung function decline and tumor growth resume when treatment is interrupted.

Sensitive and specific biomarkers of response to therapy and/or disease progression, including biomarkers of tumor metabolic activity, would facilitate clinical trials of novel therapeutic agents for LAM and enable optimization of current rapamycin-based regimens.

Our preclinical studies showed that lipogenic pathways can be detected in preclinical animal models of TSC and LAM using PET-based metabolic imaging.

The proposed study aims to quantitatively and non-invasively assess metabolic activity and response to rapamycin in LAM patients using [11C]acetate positron emission tomography (PET) imaging.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of LAM (or TSC-LAM)
* age 18 or over
* at least one renal angiomyolipoma (at least 1 cm in each diameter) confirmed by CT or MRI
* no prior treatment with rapamycin/rapalogs OR candidate for initiating treatment with rapamycin/rapalogs OR under treatment with rapamycin/rapalogs for minimum 3 months and maximum of 1 year

Exclusion Criteria:

* under treatment with rapamycin or rapalogs for < 3 months or > 1 year
* participated in research studies involving radiation exposure (> 50 mSv/year) in the past 12 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen P Priolo, MD PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seven women with Lymphangioleiomyomatosis (LAM) and at least one renal angiomyolipoma greater than 1 cm diameter were recruited to participate in the imaging study.
  Patients were recruited between August 2021 and May 2024 and signed a consent form either in person or electronically.
Pre-assignment Details: One patient became ineligible after undergoing a renal procedure.
Groups:
- Undergoing [11C]Acetate PET/CT Imaging: Patients underwent a single [11C]acetate positron emission tomography (PET)/computed tomography (CT) scan
Period: Overall Study
Arm/Group | Undergoing [11C]Acetate PET/CT Imaging
Started | 7
Completed | 6
Not Completed | 1
Not completed — One patient became ineligible after undergoing a renal procedure. | 1

BASELINE CHARACTERISTICS:
Population: One patient became ineligible after undergoing a renal procedure.
Arm/Group | Undergoing [11C]Acetate PET/CT Imaging
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants] — 18 years old or older
  Participants
    <=18 years | 0
    Between 18 and 65 years | 6
    >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Only women are affected by Lymphangioleiomyomatosis (LAM)
  Participants
    Female | 7
    Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — No race was excluded
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 1
    White | 6
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Quantitative Analysis of [11C]Acetate Uptake in LAM Lesions
Description: Standardized uptake value (SUV) will be used to quantify uptake of [11C]acetate in kidney angiomyolipoma
Time Frame: Single assessment (day of imaging)
Population: These participants had not received treatment with mTORC1 inhibitors at the time of imaging
Measure: Mean (Standard Deviation); unit: Standardized Uptake Value (SUV)
Arm/Group | Undergoing [11C]Acetate PET/CT Imaging
Number analyzed (Participants) | 4
Standardized Uptake Value (SUV) | 6.42 (3.34) [1.48 to 12.29]

2. Secondary Outcome: Quantitative Analysis of [11C]Acetate Uptake in LAM Lesions Following Treatment With mTORC1 Inhibitor
Description: Standardized uptake value (SUV) will be used to quantify uptake of [11C]acetate in kidney angiomyolipoma following treatment with mTORC1 inhibitor
Time Frame: Single assessment conducted while participants were on treatment with mTORC1 inhibitor (day of imaging)
Population: These participants were on treatment with mTORC1 inhibitor at the time of imaging
Measure: Mean (Standard Deviation); unit: Standardized Uptake Value (SUV)
Groups:
- Undergoing [11C]Acetate PET/CT Imaging: Patients underwent a single [11C]acetate positron emission tomography (PET)/computed tomography (CT) scan after treatment with mTORC1 inhibitor
Arm/Group | Undergoing [11C]Acetate PET/CT Imaging
Number analyzed (Participants) | 2
Standardized Uptake Value (SUV) | 2.80 (0.90)

ADVERSE EVENTS:
Time Frame: From imaging up to 10 days
Description: Risk of arterial catheter line (local swelling, redness, pain, infection)
Arm/Group | Undergoing [11C]Acetate PET/CT Imaging
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT05467397/Prot_SAP_002.pdf
  • Informed Consent Form (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT05467397/ICF_003.pdf